CLINICAL TRIAL: NCT04978051
Title: Randomized, Open, Multicenter Phase II Clinical Trial, Proof of Concept, to Evaluate Efficacy and Safety of Icatibant in Hospitalized Patients With SARS-COV-2 (COVID-19) Without Assisted Ventilation Compared With Standard Care
Brief Title: Investigating the Efficacy and Safety ICATIBANT For The Treatment of Patients With SARS-CoV-2 (COVID-19) Infection
Acronym: ICAT·COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sebastian Videla (Other)
Responsible Party: Sponsor-Investigator, Sebastian Videla, Head of the Clinical Research Support Unit, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-MdI-ICAT·COVID-201
Record Dates: First submitted 2021-06-30; First posted 2021-07-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia
Keywords: icatibant
MeSH Terms: interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (SoC) (Active Comparator)
  Interventions: Other: SoC
- SoC + Icatibant (Experimental)
  Interventions: Drug: Firazyr; Other: SoC

INTERVENTIONS:
Drug: Firazyr — Icatibant 10 MG/ML Prefilled Syringe
  Arms: SoC + Icatibant
Other: SoC — The SoC could include respiratory support measures, fluid therapy, antipyretic treatment, postural measures, low-molecular-weight-heparins, corticosteroids, such as dexamethasone, remdesivir and other therapeutic options

SUMMARY:
To study the efficacy and safety of icatibant in adult patients admitted to hospitalization units for pneumonia caused by COVID-19, without mechanical ventilation, 10±1 days after starting treatment or discharge from hospital if this occurs before 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (18 years or older), both sexes
2. Sars-CoV-2 infection confirmed by PCR less than 4 days before randomization
3. hospitalized with a diagnosis of SARS-CoV-2 pneumonia
4. radiographic evidence of pulmonary infiltrates
5. grade 4 or 5 on the ordinal scale for the evaluation of the patient's clinical condition
6. pO2/FiO2 <380
7. men and women of childbearing age who have heterosexual relations must be agreement to use the safe method(s) of contraception
8. obtaining the informed consent of the patient or the legal representative.

Exclusion Criteria:

1. imminent death (life expectancy less than 72h)
2. known hypersensitivity or known adverse reactions to the study drug, or its metabolites or excipients of the formulation
3. invasive mechanical ventilation
4. participation in any other clinical trial
5. ALT or AST > 5 x ULN
6. creatinine clearance <50 mL/min using the Cockcroft-Gault formula for participants '18 years old [Cockcroft 1976]
7. patients with recent acute coronary syndrome (<1 month)
8. patients with a history of stroke
9. positive pregnancy test
10. pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Efficacy of experimental treatment | up to 10 days
  Number of patients reaching grade 2 (inpatient, no longer requiring supplemental oxygen and no longer requiring care or grade 1 (hospital discharge) of the ordinal scale of the clinical state of the patient for 48 hours.
Safety of experimental treatment | up to 10 days
  Number of patients without an adverse reaction scoring 3, 4 or 5 according to the Criteria of Adverse Event Terminology (CTC-AE).

SECONDARY OUTCOMES:
Long-term efficacy | up to 10 days
  Number (percentage) of patients who reach grade 2 or grade 1 during the 10 days of to have initiated treatment.
Time to achive a clinical response | up to 40 days
  period time (days) between visit 1 (treatment start visit) and the day of gathering sustained 48-hour grade 2, grade 1 or grade 0 classification on the WHO 8-point ordinal scale for clinical status assessment The patient must be discharged from the hospital by the 28th day without a relapse or comorbidity related to COVID-19
Time to achive an afebrile state | up to 40 days
  period time (days) to reach a 48-hour sustained afebrile state (i.e., body temperature ≤ 37.5ºC) without antipyretic medication.
time from symptom onset to treatment | up to day 1
  period time (days) between the first COVID-19-related symptom and visit 1 (treatment start visit).
Responders | up to 40 days
  Number (percentage) of patients considered as responders based on National Early Warning Score 2 (NEWS 2)
COVID-19 related relapse | up to 40 days
  number (and percentage) of patients discharged who presents any COVID-19-related relapse or comorbidity
Patients with Adverse Events | up to 40 days
  number of patients with Any Adverse Events
Adverse Events | up to 40 days
  Number of Adverse Events
Serious Adverse Events | up to 40 days
  Number of Serious Adverse Events
Overall mortality | up to 40 days
  number of patients who died
COVID-19 related mortality | up to 40 days
  number of patients who died due to COVID-19
Time until death | up to 40 days
  number of days from visit 1 until death
COVID-19-related complications | up to 40 days
  number of patients who had any COVID-19 related complications
Patients requiring intensive care | up to 40 days
  number of patients who require intensive care
patients requiring intensive care and invasive mechanical ventilation | up to 40 days
  number of patients who require intensive care and invasive mechanical ventilation
patients requiring oxygen supplementation | up to 40 days
  number of patients who require oxygen supplementation from hospital discharge up until visit 7
Patients with nonsocomial infection | up to 40 days
  number (and percentage) of patients diagnosed with another nosocomial infection
Rehospitalizations | up to 40 days
  number (and percentage) of patients who requires hospital readmission within 28 (± 3) days from hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bova M, Guilarte M, Sala-Cunill A, Borrelli P, Rizzelli GM, Zanichelli A. Treatment of ACEI-related angioedema with icatibant: a case series. Intern Emerg Med. 2015 Apr;10(3):345-50. doi: 10.1007/s11739-015-1205-9. Epub 2015 Feb 10. PMID 25666515
- [Background] Busse PJ, Christiansen SC. Hereditary Angioedema. N Engl J Med. 2020 Mar 19;382(12):1136-1148. doi: 10.1056/NEJMra1808012. No abstract available. PMID 32187470
- [Background] Bygum A, Caballero T, Grumach AS, Longhurst HJ, Bouillet L, Aberer W, Zanichelli A, Botha J, Andresen I, Maurer M; IOS Study Group. Elderly versus younger patients with hereditary angioedema type I/II: patient characteristics and safety analysis from the Icatibant Outcome Survey. Clin Transl Allergy. 2019 Jul 19;9:37. doi: 10.1186/s13601-019-0272-9. eCollection 2019. PMID 31360439
- [Background] Cicardi M, Banerji A, Bracho F, Malbran A, Rosenkranz B, Riedl M, Bork K, Lumry W, Aberer W, Bier H, Bas M, Greve J, Hoffmann TK, Farkas H, Reshef A, Ritchie B, Yang W, Grabbe J, Kivity S, Kreuz W, Levy RJ, Luger T, Obtulowicz K, Schmid-Grendelmeier P, Bull C, Sitkauskiene B, Smith WB, Toubi E, Werner S, Anne S, Bjorkander J, Bouillet L, Cillari E, Hurewitz D, Jacobson KW, Katelaris CH, Maurer M, Merk H, Bernstein JA, Feighery C, Floccard B, Gleich G, Hebert J, Kaatz M, Keith P, Kirkpatrick CH, Langton D, Martin L, Pichler C, Resnick D, Wombolt D, Fernandez Romero DS, Zanichelli A, Arcoleo F, Knolle J, Kravec I, Dong L, Zimmermann J, Rosen K, Fan WT. Icatibant, a new bradykinin-receptor antagonist, in hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):532-41. doi: 10.1056/NEJMoa0906393. PMID 20818888
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Yang G, Tan Z, Zhou L, Yang M, Peng L, Liu J, Cai J, Yang R, Han J, Huang Y, He S. Effects of Angiotensin II Receptor Blockers and ACE (Angiotensin-Converting Enzyme) Inhibitors on Virus Infection, Inflammatory Status, and Clinical Outcomes in Patients With COVID-19 and Hypertension: A Single-Center Retrospective Study. Hypertension. 2020 Jul;76(1):51-58. doi: 10.1161/HYPERTENSIONAHA.120.15143. Epub 2020 Apr 29. PMID 32348166
- [Background] Hess R, Wujak L, Hesse C, Sewald K, Jonigk D, Warnecke G, Fieguth HG, de Maat S, Maas C, Bonella F, Preissner KT, Weiss B, Schaefer L, Kuebler WM, Markart P, Wygrecka M. Coagulation factor XII regulates inflammatory responses in human lungs. Thromb Haemost. 2017 Oct 5;117(10):1896-1907. doi: 10.1160/TH16-12-0904. Epub 2017 Aug 17. PMID 28816340
- [Background] Leach JK, Spencer K, Mascelli M, McCauley TG. Pharmacokinetics of single and repeat doses of icatibant. Clin Pharmacol Drug Dev. 2015 Mar;4(2):105-11. doi: 10.1002/cpdd.138. Epub 2015 Feb 2. PMID 27128215
- [Background] Siddiqi HK, Mehra MR. COVID-19 illness in native and immunosuppressed states: A clinical-therapeutic staging proposal. J Heart Lung Transplant. 2020 May;39(5):405-407. doi: 10.1016/j.healun.2020.03.012. Epub 2020 Mar 20. No abstract available. PMID 32362390
- [Background] Van De Veerdonk FL, Netea MG, van Deuren M, van der Meer JWM, de Mast Q, Brüggemann RJ, van der Hoeven H. Kinins and cytokines in COVID-19: a comprehensive pathophysiological approach. 10.20944/preprints202004.0023.v1.
- [Background] Jin YH, Cai L, Cheng ZS, Cheng H, Deng T, Fan YP, Fang C, Huang D, Huang LQ, Huang Q, Han Y, Hu B, Hu F, Li BH, Li YR, Liang K, Lin LK, Luo LS, Ma J, Ma LL, Peng ZY, Pan YB, Pan ZY, Ren XQ, Sun HM, Wang Y, Wang YY, Weng H, Wei CJ, Wu DF, Xia J, Xiong Y, Xu HB, Yao XM, Yuan YF, Ye TS, Zhang XC, Zhang YW, Zhang YG, Zhang HM, Zhao Y, Zhao MJ, Zi H, Zeng XT, Wang YY, Wang XH; , for the Zhongnan Hospital of Wuhan University Novel Coronavirus Management and Research Team, Evidence-Based Medicine Chapter of China International Exchange and Promotive Association for Medical and Health Care (CPAM). A rapid advice guideline for the diagnosis and treatment of 2019 novel coronavirus (2019-nCoV) infected pneumonia (standard version). Mil Med Res. 2020 Feb 6;7(1):4. doi: 10.1186/s40779-020-0233-6. PMID 32029004
- [Background] Zanichelli A, Maurer M, Aberer W, Caballero T, Longhurst HJ, Bouillet L, Fabien V, Andresen I; IOS Study Group. Long-term safety of icatibant treatment of patients with angioedema in real-world clinical practice. Allergy. 2017 Jun;72(6):994-998. doi: 10.1111/all.13103. Epub 2017 Mar 13. PMID 27926986
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Derived] Malchair P, Giol J, Garcia V, Rodriguez O, Ruibal JC, Zarauza A, Llopis F, Matellan L, Bernal T, Solis B, Otero A, Carnaval T, Jofre H, Jacob J, Solanich X, Antoli A, Rocamora G, Videla S. Three-Day Icatibant on Top of Standard Care in Patients With Coronavirus Disease 2019 Pneumonia: A Randomized, Open-Label, Phase 2, Proof-of-Concept Trial. Clin Infect Dis. 2023 May 24;76(10):1784-1792. doi: 10.1093/cid/ciac984. PMID 36610464
- [Derived] Malchair P, Otero A, Giol J, Solanich X, Carnaval T, Fernandez-Nistal A, Sanchez-Gabriel A, Montoto C, Lleonart R, Videla S; ICAT-COVID team. A multicenter, open-label, randomized, proof-of-concept phase II clinical trial to assess the efficacy and safety of icatibant in patients infected with SARS-CoV-2 (COVID-19) and admitted to hospital units without invasive mechanical ventilation: study protocol (ICAT-COVID). Trials. 2022 Apr 12;23(1):303. doi: 10.1186/s13063-022-06219-7. PMID 35413921
- See also: COVID19, WHO — http://covid19.who.int.
- See also: Icatibant (Firazyr®). Ficha técnica, Febrero 2019. — https://cima.aemps.es/cima/pdfs/es/ft/08461001/FT_08461001.pdf